CLINICAL TRIAL: NCT00393653
Title: Prescription Methods Assessment Project (PMAP)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended early
Sponsor: American Academy of Family Physicians (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 06-016
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Osteoarthritis; Gastroesophageal Reflux Disease
Keywords: osteoarthritis; gastroesophageal reflux disease; practice-based research; N-of-1 trial; prescription; single-patient trial
MeSH Terms: conditions — Osteoarthritis; Gastroesophageal Reflux

INTERVENTIONS:
Procedure: N-of-1 prescription method

SUMMARY:
The purpose of this study is to evaluate whether a novel prescription method (N-of-1 intervention)can be successfully integrated into primary care practices and to examine the effects of this prescription method on selected patient health outcomes (e.g.., medication compliance, medication costs, symptom management, satisfaction of physician/patient visit, etc.) in patients with a uncontrolled or new diagnosis of Osteoarthritis or Chronic Heartburn (GERD).

DETAILED DESCRIPTION:
The current prescription writing behavior of physicians is largely an informed decision based upon education and experience. The physician typically assesses the signs and symptoms of a patient presentation, laboratory and other clinical tests, and other factors that may be known to the physician (e.g. an inability to swallow capsules, or a requirement to be in direct sunlight for an extended period), and chooses a drug to prescribe with no evidence of patient response to the agent prescribed. The prescribing physician may or may not decide to validate this decision by additional testing in the form of follow-up visits or other procedures that are designed to assess the effectiveness of the prescription after some arbitrary period of time, but not comparatively with other available agents.

Other influences may impact the decision including aggressive promotions by pharmaceutical companies in support of their latest medication and direct to consumer retail advertising. Studies conducted by the University of Washington Medical School have shown that when patients merely enquire about a drug for which they've seen advertising, that drug is then more frequently prescribed (Hollon 2005). At its best, prescription writing is an educated guess with a scheduled follow-up to verify the results of the decision. At its worst, it may result in all risk with no benefit to the patient if the patient is a non-responder, or if the patient accepts an adverse outcome without informing the physician.

The Opt-e-scrip method for determining prescriptions is virtually the same method that is used to assess new drugs for regulatory approval (i.e.,controlled experiments to reduce systematic error, reduce random variation, increase precision of assessment). However, instead of applying the techniques of scientific investigation to populations, these methods are applied to the individual patient. Opt-e-scrip's proprietary methods are used to assess alternative choices within a therapeutic class for effectiveness and safety before prescribing a specific agent for an individual patient. In this case, however, because the drugs are already marketed and cost information is available, when two or more agents are equally safe and effective, a decision can be made reliably on cost as a relevant factor (2006).

Initial studies indicate that the Opt-e-scrip methodology can distinguish between similar medications based on efficacy and/or side effects at the individual patient level in patients with osteoarthritis, gastroesophageal reflux disease (GERD), and allergic rhinitis (Reitberg, Del Rio et al. 2002; Reitberg, Weiss et al. 2005). It remains to be seen how well this method can be integrated into clinical care and how clinicians and patients respond to the method as part of routine care. This project will assess the integration of Opt-e-scrip method into 20 primary care practices that will each use the method to assist with medication selection in 30 to 40 patients with a new diagnosis or uncontrolled osteoarthritis and GERD.

Specific Aims of Study.

* 1. Evaluate whether the (N-of-1) intervention prescription method can be successfully integrated into primary care practices.
* 2. Determine whether use of the intervention prescription method changes medication selection for patients with osteoarthritis and gastroesophageal reflux disease.
* 3. Examine the effects of the intervention method on medication compliance.
* 4. Examine the effects of the intervention prescription method on medication costs.

References

1. Hollon, M. F. (2005). "Direct-to-consumer advertising: a haphazard approach to health promotion." Jama 293(16): 2030-3.
2. Opt-e-scrip, I. (2006). Optimizing each prescription to the individual, Opt-e-scrip. 2006.
3. Reitberg, D. P., E. Del Rio, et al. (2002). "Single-patient drug trial methodology for allergic rhinitis." Ann Pharmacother 36(9): 1366-74.
4. Reitberg, D. P., S. L. Weiss, et al. (2005). "Advances in Single-Patient Trials for Drug Treatment Optimization and Risk Management." Drug Information Journal 39: 119-124.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* capable of giving informed consent
* a new diagnosis or uncontrolled symptoms of either osteoarthritis or gastroesophageal reflux disease
* if new diagnosis or uncontrolled osteoarthritis, patient must have condition in knee or hip (need not be isolated)

Exclusion Criteria:

* too ill to participate
* not capable of giving informed consent
* not able to be contacted via phone for study follow-up
* unable to read English, including blindness
* if treating physician considers patient to have medical conditions that would cause the patient to be placed at risk by trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2006-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Side-effects and adverse events (base-line, 3 and 6 months)

SECONDARY OUTCOMES:
Symptoms of condition and health related issues (i.e., satisfaction of doctor visit, self-efficacy)at baseline, 3 and 6 months
Patient medication information and adherence to prescription(s) at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wilson D Pace, MD, Principal Investigator — American Academy of Family Physicians
Locations (1):
- American Academy of Family Physicians National Research Network, Leawood, Kansas, United States

REFERENCES:
- [Background] Wolfe B, Del Rio E, Weiss SL, Mendelson A, Elbaga TA, Huser FJ, Reitberg DP. Validation of a single-patient drug trial methodology for personalized management of gastroesophageal reflux disease. J Manag Care Pharm. 2002 Nov-Dec;8(6):459-68. doi: 10.18553/jmcp.2002.8.6.459. PMID 14613380
- [Background] Reitberg DP, Del Rio E, Weiss SL, Rebell G, Zaias N. Single-patient drug trial methodology for allergic rhinitis. Ann Pharmacother. 2002 Sep;36(9):1366-74. doi: 10.1345/aph.1C031. PMID 12196053